CLINICAL TRIAL: NCT02039466
Title: The Effect of Pressure-controlled Ventilation on the Respiratory Complication in Patients Undergoing Laparoscopic Colectomy Compared With Volume-controlled Ventilation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, So Young Yang, So Young Yang. MD.PHD, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ChungAng UH
Record Dates: First submitted 2014-01-16; First posted 2014-01-17 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Postoperative Respiratory Complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- volume controlled ventilation (Active Comparator): volume controlled ventilation as a tidal volume of 8 ml/kg (ideal body weight)
  Interventions: Procedure: volume controlled ventilation
- pressure controlled ventilation (Active Comparator): pressure controlled ventilation as a tidal volume of 8 ml/kg (ideal body weight)
  Interventions: Procedure: pressure controlled ventilation

INTERVENTIONS:
Procedure: volume controlled ventilation
  Arms: volume controlled ventilation
Procedure: pressure controlled ventilation
  Arms: pressure controlled ventilation

SUMMARY:
Postoperative pulmonary complications following abdominal surgery are frequent and associated with increased morbidity and mortality and hospital length of stay. Pressure controlled ventilation will improve oxygenation indices , hemodynamics during anesthesia for laparoscopic colectomy, decreasing postoperative pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status classification
* patients scheduled for laparoscopic colectomy

Exclusion Criteria:

* severe cardiopulmonary disease
* patients who cannot understand Korean

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
peak airway pressure in patients receiving pressure controlled ventilation and volume controlled ventilation | 40 minutes after pneumoperitoneum

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Hospital, Seoul, Seoul, South Korea